CLINICAL TRIAL: NCT02795598
Title: Diaphragmatic Dysfunction After Ultrasound-guided Supraclavicular Brachial Plexus Block With Single or Double Injection Technique
Brief Title: Diaphragmatic Dysfunction After Ultrasound-guided Supraclavicular Block With Single or Double Injection Technique
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study protocol changed significantly and a new file was started.
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1021191
Record Dates: First submitted 2016-05-27; First posted 2016-06-10 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2016-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single Injection Supraclavicular Block (Active Comparator): Patients scheduled for surgery distal to the elbow will have an ultrasound guided single injection supraclavicular nerve block for surgical anesthesia.
  Interventions: Procedure: Single injection supraclavicular nerve block
- Double Injection Supraclavicular Block (Active Comparator): Patients scheduled for surgery distal to the elbow will have an ultrasound guided double injection supraclavicular nerve block for surgical anesthesia.
  Interventions: Procedure: Double injection supraclavicular nerve block

INTERVENTIONS:
Procedure: Single injection supraclavicular nerve block — The ultrasound probe will be applied in a sterile fashion in the supraclavicular fossa to obtain a short-axis view of the subclavian artery. A 22G, 50mm Echogenic Stimuplex needle will be advanced in-plane with respect to the image, and the needle tip will be advanced to the junction of the first rib and subclavian artery. Ultrasound cineloops will be kept of all nerve block procedures.
  30 milliliters of mepivacaine 1.5% will be injected incrementally in 5ml boluses at this location looking for spread of local anesthetic under and medial to the subclavian artery. The needle may be slightly repositioned to improve the distribution of the injectate at the discretion of the attending anesthesiologist.
  Arms: Single Injection Supraclavicular Block
Procedure: Double injection supraclavicular nerve block — The ultrasound probe will be applied in a sterile fashion in the supraclavicular fossa to obtain a short-axis view of the subclavian artery. A 22G, 50mm Echogenic Stimuplex needle will be advanced in-plane with respect to the image, and the needle tip will be advanced to the junction of the first rib and subclavian artery. Ultrasound cineloops will be kept of all nerve block procedures.
  15 milliliters of mepivacaine 1.5% will be injected incrementally at the same, above-mentioned location. The needle will then be redirected to the superolateral aspect of the brachial plexus, and an additional 15ml will be injected here. Again, the needle may slightly repositioned at the discretion of the attending anesthesiologist in order to obtain adequate spread.
  Arms: Double Injection Supraclavicular Block

SUMMARY:
The investigators plan to determine the incidence of hemi-diaphragmatic paresis (HDP) with two commonly used techniques of supraclavicular nerve block, the single and double injection techniques.

It is our hypothesis that a double injection peripheral nerve block technique will increase the risk of HDP when compared to a single injection technique.

DETAILED DESCRIPTION:
The investigators will perform a prospective, blinded, randomized controlled trial to assess the two methods of supraclavicular block (single and double injection), and the resultant incidence of temporary diaphragm dysfunction, or hemi-diaphragmatic paresis (HDP) will be measured with ultrasound. Patients having forearm or hand surgery will be asked by the attending anesthesiologist if they will agree to be approached by someone from the research team for consent and possible inclusion in the study. This will be done in the anesthesia preoperative assessment clinic, or in the pre-op area on the day of surgery (if a patient was not seen in clinic).

Once consented, all patients in the study will have baseline measurements of their sensation and movement of the arm for surgery, as well as an ultrasound examination of the movement of the diaphragm.

Patients will then be randomized to either the single or double injection supraclavicular nerve block. The blocks will be performed by attending anesthesiologists with experience in regional anesthesia, or by residents and fellows under the direct supervision of such anesthesiologists.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for unilateral upper extremity surgery below the level of the elbow (the forearm or hand) who are having a regional block for anesthesia
* Patient must be over 18 years old
* Weight greater than 50kg
* English speaking
* Be available to be contacted by phone on post-operative day 1
* ASA physical status 1-3
* BMI under 35 kg/m2

Exclusion Criteria:

* Inability to consent to study participation
* Pre-existing neuromuscular disease or severe neurological dysfunction
* Severe coagulopathy
* Severe obstructive or restrictive lung disease
* Pregnancy
* Prior surgery in the supraclavicular region
* Allergy to medications used in the study
* Known diaphragmatic dysfunction of either diaphragm
* Inability to visualize the diaphragm with ultrasound on the side of the surgical procedure
* Highly opioid-tolerant patient (>40mg of morphine PO or equivalent per day for >1month)
* Patient requests a general anesthesia technique
* Attending anesthesiologist preference for alternate anesthetic technique
* Surgeon or attending anesthesiologist request for a different anesthesia technique
* Current involvement in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Hemidiaphragmatic paresis (HDP) by diaphragmatic thickening | Relative change in ultrasound assessment of diaphragmatic thickening (Baseline vs 30 min after supraclavicular block)
  Ultrasound measurement of diaphragmatic thickening

SECONDARY OUTCOMES:
Onset time of sensory block | Baseline, 5, 10, 15, 20, 25, and 30 minutes after block
  Sensation of the terminal peripheral nerves of the upper extremity will be assessed by a single observer blinded to the technique for the musculocutaneous, median, radial, ulnar and the medial antebrachial cutaneous nerves. Sensory assessments will be done using a blunt needle and the response will be assessed on a 3-point scale using the contralateral limb as a control: 0 = normal sensation, 1 = hypoesthesia, and 2 = anesthesia. A composite score will be created for each time point.
Onset time of motor block | Baseline, 5, 10, 15, 20, 25, and 30 minutes after block
  Motor blockade of the musculocutaneous, radial, median, and ulnar nerves will be evaluated by elbow flexion, thumb abduction, thumb opposition, and thumb adduction, respectively. Motor blockade will be graded on a 3-point scale: 0 = normal strength, 1 = weakness relative to the contralateral side, and 2 = complete paralysis. A composite score will be created for each time point.
Bedside spirometry - forced expiratory volume at one second (FEV1) | Relative change in FEV1 (Baseline vs 30 min after supraclavicular block)
  Relative changes in forced expiratory volume at one second (FEV1) will be compared
Bedside spirometry - forced vital capacity (FVC) | Relative change in FVC (Baseline vs 30 min after supraclavicular block)
  Relative changes in forced vital capacity (FVC) will be compared
Dyspnea | 30 minutes after the supraclavicular block
  Patient will be asked if they are having shortness of breath.
Procedure performance time | From the time that the block needle enters skin until it is removed
  Measurement of time taken to perform both types of block
Incidence of complications | From block performance until 24 hours after block is completed (24 hour follow-up call)
  The incidence of complications, including puncturing a vessel, or post-operative sensory or movement problems
Clinical Efficacy | At the time of surgery start
  Nerve blocks will be considered clinically efficacious if surgery is able to proceed without the need for additional local anesthesia at the site or need for general anesthesia. Any use of supplemental local or general anesthesia will be considered a block failure.
Incidence of Hemidiaphragmatic paresis (HDP) by diaphragmatic excursion | Relative change in ultrasound assessment of diaphragmatic excursion (Baseline vs 30 min after supraclavicular block)
  Ultrasound measurement of HDP

CONTACTS AND LOCATIONS:
Overall Officials: Kwesi Kwofie, MD, Principal Investigator — Nova Scotia Health Authority

IPD SHARING:
Plan to Share IPD: Undecided